CLINICAL TRIAL: NCT06848322
Title: The Effects of 8-week Resistance and Aerobic Exercise on Anxiety, Depression, Sleep, Inhibitory Control in Young Adults With Smartphone Overdependence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seoul (Other)
Responsible Party: Principal Investigator, Hyeongchan Lee, University of Seoul, University of Seoul
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UOS 2024-08-007-004
Record Dates: First submitted 2025-02-09; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Exercise; Smartphone Addiction; Sleep; Inhibition; Mood
MeSH Terms: conditions — Motor Activity; Internet Addiction Disorder; Inhibition, Psychological | interventions — Resistance Training; Exercise

STUDY DESIGN:
Intervention Model Description: resistance exercise group → Experimental aerobic exercise group → Experimental control → No Intervention There are three groups in this study: the resistance exercise group, the aerobic exercise group, and the control group. Measurements are conducted at three time points: pre-intervention, mid-intervention (4 weeks after the intervention), and post-intervention
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- resistance exercise group (Experimental): They will perform resistance exercise for 8 weeks.
  Interventions: Behavioral: resistance exercise
- aerobic exercise group (Experimental): They will perform aerobic exercise for 8 weeks.
  Interventions: Behavioral: aerobic exercise
- control group (Sham Comparator): They will maintain their usual lifestyle for 8 weeks.
  Interventions: Other: Control (placebo)

INTERVENTIONS:
Behavioral: resistance exercise — Participants will perform resistance exercise for 8 weeks
  Other Names: aerobic exercise; control
  Arms: resistance exercise group
Behavioral: aerobic exercise — Participants will perform aerobic exercise for 8 weeks
  Arms: aerobic exercise group
Other: Control (placebo) — Participants will maintain their usual lifestyle for 8 weeks.
  Arms: control group

SUMMARY:
The purpose of this study is to identify the effects of the resistance exercise and aerobic exercise on depression, anxiety, sleep, inhibitory control in young adult with smartphone overdependence

ELIGIBILITY:
Inclusion Criteria:

* Smartphone overdependent scale score of 24 ≥
* No regular exercise in the past 3 months

Exclusion Criteria:

* Unable to perform exercise
* Patients with musculoskeletal disorders
* Patients with cardiovascular diseases.

Ages: 20 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-05 (Actual)

PRIMARY OUTCOMES:
sleep duration | pre intervention: for 8days(before the intervention) / post intervention: for 8days(after the intervention)
  In this study, we will assess participants' sleep duration using a wrist-worn GENEActiv triaxial accelerometer (Activinsights, Cambridge, UK). Participants will be instructed to wear the device on their non-dominant wrist 24 hours a day for 8 days, except during contact sports that may pose a risk of injury. Sleep duration (minutes) is defined as the total time spent sleeping.
Sleep efficiency | pre intervention: for 8days(before the intervention) / post intervention: for 8days(after the intervention)
  In this study, we will assess participants' sleep efficiency using a wrist-worn GENEActiv triaxial accelerometer (Activinsights, Cambridge, UK). Participants will be instructed to wear the device on their non-dominant wrist 24 hours a day for 8 days, except during contact sports that may pose a risk of injury. Sleep efficiency(%) is defined as the proportion of time spent asleep relative to time in bed
Time in bed | pre intervention: for 8days(before the intervention) / post intervention: for 8days(after the intervention)
  In this study, we will assess participants' time in bed using a wrist-worn GENEActiv triaxial accelerometer (Activinsights, Cambridge, UK). Participants will be instructed to wear the device on their non-dominant wrist 24 hours a day for 8 days, except during contact sports that may pose a risk of injury. Time in bed (minutes) is defined as the total time spent in bed, including both sleep and wakefulness
Sleep onset time | pre intervention: for 8days(before the intervention) / post intervention: for 8days(after the intervention)
  In this study, we will assess participants' sleep onset time using a wrist-worn GENEActiv triaxial accelerometer (Activinsights, Cambridge, UK). Participants will be instructed to wear the device on their non-dominant wrist 24 hours a day for 8 days, except during contact sports that may pose a risk of injury. Sleep onset time (hours and minutes) is defined as the time at which sleep begins.
wake time | pre intervention: for 8days(before the intervention) / post intervention: for 8days(after the intervention)
  In this study, we will assess participants' sleep onset time using a wrist-worn GENEActiv triaxial accelerometer (Activinsights, Cambridge, UK). Participants will be instructed to wear the device on their non-dominant wrist 24 hours a day for 8 days, except during contact sports that may pose a risk of injury. Wake time (hours and minutes) is defined as the final wake-up time.

SECONDARY OUTCOMES:
Depression | pre intervention(day 1), post intervention(day 57)
  Participants will visit the laboratory to complete the Beck Depression Inventory(BDI), a self-reported questionnaire assessing depressive symptoms. The BDI consists of 21 items, each scored on a scale from 0 to 3, with total scores ranging from 0 to 63. Higher scores indicate more severe depressive symptoms
Anxiety | pre intervention(day 1), post intervention(day 57)
  Participants will visit the laboratory to complete the Beck Anxiety Inventory (BAI), a self-reported questionnaire assessing anxiety symptoms. The BAI consists of 21 items, each scored on a scale from 0 to 3, with total scores ranging from 0 to 63. Higher scores indicate more severe anxiety symptoms.
Inhibition | pre intervention(day 1), post intervention(day 57)
  The Go/NoGo task will be used to measure the inhibition The measured variables will include reaction time (RT) and accuracy.
  At the beginning of the test, a series of stimulus characters will be presented in the center of the screen one by one. Each stimulus character will be displayed for 400 ms, with a random interval of 400-700 ms between stimuli.
  Before the test, participants will be informed that "L" is a Go stimulus and "C" is a NoGo stimulus. When "L" appears in the center of the screen, participants will be required to press the space bar key with their index finger as quickly and accurately as possible. When "C" appears, participants must not respond.
  The system will record the reaction time and accuracy for Go stimuli and the accuracy for NoGo stimuli. The total number of stimulus characters will be 240, consisting of 180 Go stimuli (75%) and 60 NoGo stimuli (25%).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Seoul, Centennial Memorial Hall., Dongdaemun, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol, Informed Consent Form (ICF)
Supporting Information: Study Protocol, ICF
Time Frame: 2025.03.01~2026.03.01